CLINICAL TRIAL: NCT02186743
Title: Irritable Bowel Syndrome and Food Sensitivity: Assessing Clinical Outcomes and Inflammatory Cellular Pathways
Brief Title: Irritable Bowel Syndrome and Food Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Cell Science Systems, Corp. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1404013784
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2016-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; IBS; Diet; Food sensitivity
MeSH Terms: conditions — Irritable Bowel Syndrome; Food Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Diet (Experimental): Personalized dietary advice based on a commercially available blood test. Participants will be instructed to avoid eating selected foods for the duration of the intervention period (4 weeks). Some foods will be acceptable to consume every four days in rotation diet fashion.
  Interventions: Other: Personalized Dietary Advice
- Active control diet (Active Comparator): Personalized dietary advice based on a commercially available blood test. Participants will be instructed to avoid eating selected foods for the duration of the intervention period (4 weeks). Some foods will be acceptable to consume every four days in rotation diet fashion.
  Interventions: Other: Personalized Dietary Advice

INTERVENTIONS:
Other: Personalized Dietary Advice — Personalized dietary advice based on a commercially available blood test. Participants will be instructed to avoid eating selected foods for the duration of the intervention period (4 weeks). Some foods will be acceptable to consume every four days in rotation diet fashion.

SUMMARY:
The primary objective of the clinical trial portion of this study is to assess whether an individualized dietary plan based on a commercial food sensitivity assay provides specific benefit in a randomized controlled trial in adults with irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
This is a parallel group, randomized control trial, powered to assess changes in validated outcomes in adult patients with symptomatic irritable bowel syndrome. Subjects will receive dietary counseling and be asked to adhere to dietary instructions for 4 weeks. Assessments will occur at baseline, 4-weeks, and 8-weeks post-baseline.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-70 years of age.
* Irritable Bowel Syndrome by Rome III criteria.
* Stable dose (30 days) of concurrent IBS medications
* Agree not to make significant changes to their diet during the study
* IBS-SSS score of >150

Exclusion Criteria:

* History of major abdominal surgeries
* History of inflammatory bowel disease
* Antibiotic use within 1 month of enrollment
* Radiation proctitis or other known poorly controlled medical conditions that could interfere with bowel function
* Current use of opioid pain medications (except for NSAIDs)
* Previous experience participating in dietary studies for IBS
* Current use of medications which are known to be affected by modest dietary changes
* Vitamin C use of >2000 mg/day
* Quercetin use of >500 mg/day

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Global Improvement Scale (IBS-GIS) | Baseline
  The IBS-GIS is a single item assessment of overall IBS symptoms. It poses the question to study participants "Compared to the way you felt before you entered the study, have your IBS symptoms over the past 7 days been:" Subjects respond on a scale of 1-7 where: 1 = Substantially Worse, 2 = Moderately Worse, 3 = Slightly Worse, 4 = No Change, 5 = Slightly Improved, 6 = Moderately Improved, 7 = Substantially Improved.
Irritable Bowel Syndrome Global Improvement Scale (IBS-GIS) | 4 weeks
  The IBS-GIS is a single item assessment of overall IBS symptoms. It poses the question to study participants "Compared to the way you felt before you entered the study, have your IBS symptoms over the past 7 days been:" Subjects respond on a scale of 1-7 where: 1 = Substantially Worse, 2 = Moderately Worse, 3 = Slightly Worse, 4 = No Change, 5 = Slightly Improved, 6 = Moderately Improved, 7 = Substantially Improved.
Irritable Bowel Syndrome Global Improvement Scale (IBS-GIS) | 8 weeks
  The IBS-GIS is a single item assessment of overall IBS symptoms. It poses the question to study participants "Compared to the way you felt before you entered the study, have your IBS symptoms over the past 7 days been:" Subjects respond on a scale of 1-7 where: 1 = Substantially Worse, 2 = Moderately Worse, 3 = Slightly Worse, 4 = No Change, 5 = Slightly Improved, 6 = Moderately Improved, 7 = Substantially Improved.

SECONDARY OUTCOMES:
Irritable Bowel Syndrome Adequate Relief (IBS-AR) | Baseline
  The IBS-AR is a single item assessment of IBS symptom relief. It poses the question to study participants "Over the past week have you had adequate relief of your IBS symptoms?" Subjects respond either "yes" or "no."
Irritable Bowel Syndrome Adequate Relief (IBS-AR) | 4 weeks
  The IBS-AR is a single item assessment of IBS symptom relief. It poses the question to study participants "Over the past week have you had adequate relief of your IBS symptoms?" Subjects respond either "yes" or "no."
Irritable Bowel Syndrome Adequate Relief (IBS-AR) | 8 weeks
  The IBS-AR is a single item assessment of IBS symptom relief. It poses the question to study participants "Over the past week have you had adequate relief of your IBS symptoms?" Subjects respond either "yes" or "no."
Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS) | Baseline
  The IBS-SSS contains five questions that assess the severity of abdominal pain, the frequency of abdominal pain, the severity of abdominal distention, dissatisfaction with bowel habits, and interference with quality of life.
Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS) | 4 weeks
  The IBS-SSS contains five questions that assess the severity of abdominal pain, the frequency of abdominal pain, the severity of abdominal distention, dissatisfaction with bowel habits, and interference with quality of life.
Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS) | 8 weeks
  The IBS-SSS contains five questions that assess the severity of abdominal pain, the frequency of abdominal pain, the severity of abdominal distention, dissatisfaction with bowel habits, and interference with quality of life.
Irritable Bowel Syndrome Quality of Life Questionnaire (IBS-QoL) | Baseline
  The IBS-QoL is a 34-item measure assessing the degree to which IBS interferes with patient quality of life. Each item is rated on a 5-point Likert scale and a linear transformation yields a summed score with a theoretical range of 0 to 100, with a higher score indicating better quality of life.
Irritable Bowel Syndrome Quality of Life Questionnaire (IBS-QoL) | 4 weeks
  The IBS-QoL is a 34-item measure assessing the degree to which IBS interferes with patient quality of life. Each item is rated on a 5-point Likert scale and a linear transformation yields a summed score with a theoretical range of 0 to 100, with a higher score indicating better quality of life.
Irritable Bowel Syndrome Quality of Life Questionnaire (IBS-QoL) | 8 weeks
  The IBS-QoL is a 34-item measure assessing the degree to which IBS interferes with patient quality of life. Each item is rated on a 5-point Likert scale and a linear transformation yields a summed score with a theoretical range of 0 to 100, with a higher score indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ather Ali, ND, MPH, MHS, Principal Investigator — Yale University; Wajahat Mehal, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Result] Ali A, Weiss TR, McKee D, Scherban A, Khan S, Fields MR, Apollo D, Mehal WZ. Efficacy of individualised diets in patients with irritable bowel syndrome: a randomised controlled trial. BMJ Open Gastroenterol. 2017 Sep 20;4(1):e000164. doi: 10.1136/bmjgast-2017-000164. eCollection 2017. PMID 29018540
- See also: BMJ Open Gastroenterology — http://bmjopengastro.bmj.com/content/4/1/e000164